CLINICAL TRIAL: NCT03212131
Title: Investigation of Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Multiple Doses of Somapacitan in Subjects With Mild and Moderate Degrees of Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4298; U1111-1187-9247 (Other: World Health Organization (WHO)); 2016-003911-36 (Registry Identifier: EudraCT)
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency; Growth Hormone Deficiency in Children
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan

STUDY DESIGN:
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Normal hepatic function (Experimental): Subjects with normal hepatic function
  Interventions: Drug: Somapacitan
- Mild hepatic impairment (Experimental): Subjects with mild hepatic impairment
  Interventions: Drug: Somapacitan
- Moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — 3 once-weekly subcutaneous administrations (s.c., under the skin) of somapacitan with a dose of 0.08 mg/kg

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the effect of abnormal liver (hepatic) function on the amount of trial drug getting into the body and removal of the drug from the body (this is called pharmacokinetics).

In this trial the participants will receive three subcutaneous (under the skin) injections of the trial drug somapacitan. Somapacitan is a long-acting growth hormone analogue (a drug similar to human growth hormone) intended for once-weekly subcutaneous administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75 years (both inclusive)
* Body mass index of 18.5-39.9 kg/sqm (both inclusive)
* Subjects with normal hepatic function or hepatic impairment (mild or moderate)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice) for at least 16 days after the last trial product administration
* Male of reproductive age who or whose partner(s) is not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice) or male who is not willing to refrain from donating semen for at least 16 days after last trial product administration
* Any blood draw in excess of 25 mL in the past 30 days, or donation of blood or plasma in excess of 400 mL within the 90 days preceding screening
* Any disorder, except for conditions associated with hepatic impairment in the group of subjects with compromised hepatic function, which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
Area under the somapacitan serum concentration time curve | From time 0 to 168 hours after the last dosing on Day 15
  Calculated based on somapacitan measured in blood

SECONDARY OUTCOMES:
Maximum serum concentration of somapacitan | After the last dosing on Day 15 until Day 43
  Calculated based on plasma somapacitan activity measured in blood
Time to maximum serum concentration of somapacitan | After the last dosing on Day 15 until Day 43
  Calculated based on plasma somapacitan activity measured in blood
Incidence of adverse events | From first dosing to Day 43
  Count
Occurrence of anti-somapacitan antibodies | From Day 0 to Day 43
  Count

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Bentz Damholt B, Dombernowsky SL, Dahl Bendtsen M, Bisgaard C, Hojby Rasmussen M. Effect of Kidney or Hepatic Impairment on the Pharmacokinetics and Pharmacodynamics of Somapacitan: Two Open-Label, Parallel-Group Trials. Clin Pharmacokinet. 2021 Aug;60(8):1015-1027. doi: 10.1007/s40262-021-00990-7. Epub 2021 Mar 23. PMID 33754315